CLINICAL TRIAL: NCT02072434
Title: A Prospective, Randomized, Open-Label Blinded Endpoint Evaluation (PROBE) Parallel Group Study Comparing Edoxaban (DU-176b) With Enoxaparin/Warfarin Followed by Warfarin Alone in Subjects Undergoing Planned Electrical Cardioversion of Nonvalvular Atrial Fibrillation
Brief Title: Edoxaban vs. Warfarin in Subjects Undergoing Cardioversion of Nonvalvular Atrial Fibrillation (NVAF)
Acronym: ENSURE-AF
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DU176b-F-E308; 2013-003148-21 (EudraCT Number)
Record Dates: First submitted 2014-02-20; First posted 2014-02-26 (Estimated); Results first posted 2019-03-13 (Actual); Last update posted 2019-03-15 (Actual); Status verified 2019-03

CONDITIONS: Atrial Fibrillation
Keywords: Nonvalvular atrial fibrillation (NVAF); anti-coagulant; warfarin; edoxaban; electrical cardioversion
MeSH Terms: conditions — Atrial Fibrillation | interventions — edoxaban; Warfarin; Enoxaparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Edoxaban (Experimental): Edoxaban oral tablet, 60 mg-once daily (QD), reduced to 30 mg based on protocol-defined parameters, for up to 49 days
  Interventions: Drug: Edoxaban
- Warfarin (Active Comparator): Participants naïve to anticoagulation, taking anticoagulants other than a Vitamin K antagonist (VKA) or taking a VKA but with a prothrombin time (PT) international normalized ratio (INR) of less than 2.0 receive enoxaparin until they reach a PT INR of at least 2.0, before taking warfarin.
  All participants in this arm receive warfarin oral tablet QD at their doctor's prescribed dose, for up to 49 days.
  Interventions: Drug: Warfarin; Drug: Enoxaparin

INTERVENTIONS:
Drug: Edoxaban — Edoxaban 30 mg tablets for oral administration
  Arms: Edoxaban
Drug: Warfarin — Warfarin tablet, 1.0 or 2.5 mg, for oral administration
  Arms: Warfarin
Drug: Enoxaparin — Enoxaparin per label, at prescribed dose until PT INR at least 2.0
  Arms: Warfarin

SUMMARY:
The purpose of this study is to compare edoxaban to warfarin (with enoxaparin, if needed). It will see if edoxaban prevents stroke and other blood clotting problems as well and as safely as warfarin. People with atrial fibrillation (irregular heartbeat) might be able to join. Their doctors must plan to use shock to make their hearts beat normally. About 2200 people from different countries will join. They will have an equal chance of receiving either treatment. They are anticipated to be in the study for around 82 days. Tests will include physicals and finger-pricks. Participants will provide blood and urine samples.

DETAILED DESCRIPTION:
The purpose of this study is to compare edoxaban (investigational drug) with warfarin and enoxaparin, to see if it is safe and effective in preventing stroke and other blood clot complications in subjects with atrial fibrillation whose doctors plan to treat them with an electrical cardioversion. It is expected that 284 sites will recruit 2200 subjects from North America, EU, Russia, Ukraine and Israel. Participants will be randomly allocated to receive either treatment with edoxaban, or treatment with warfarin, plus enoxaparin if required. Participants will have an equal chance of receiving either treatment. Participants will be in the study for a maximum of 82 days. Study procedures will include physical examinations, vital signs (pulse and sitting blood pressure), ECG (electrocardiogram), finger prick blood clotting tests, blood samples and urine samples.

The study is expected to show that edoxaban will provide comparable incidence rates to warfarin plus enoxaparin, the current standard treatment for both efficacy and bleeding.

ELIGIBILITY:
Inclusion Criteria:

* Has signed informed consent
* Is older than minimum legal adult age (country specific)
* Has had ongoing AF lasting at least 48 hrs but <= 12 months (with or without valvular heart disease)
* Has treatment plan that includes for electrical cardioversion
* Has NVAF or other specific valvular heart diseases (eg, mitral valve prolapse, mitral valve regurgitation, and aortic valve disease)

Exclusion Criteria:

* Has AF that is transient or reversible
* Has contraindicated condition, ie, conditions considered to be formal indication for conventional anticoagulation
* Has a history of left atrial appendage (LAA) closure
* Has a known thrombus in LAA, the left atrial, left ventricle or aorta - or an intracardial mass
* Has had myocardial infarction (MI), stroke, acute coronary syndrome (ACS), or percutaneous coronary intervention (PCI) within the past 30 days
* Has any contraindication to anticoagulant agents
* Has had protocol-defined signs of bleeding or conditions associated with high risk of bleeding that would preclude participation
* Is receiving, or plans to receive during the study period, dual antiplatelet therapy (DAPT) or invasive procedures (other than routine endoscopy) in which bleeding would be anticipated
* Has received prohibited concomitant medication or therapy
* Has had protocol-defined signs of bleeding or high
* Has inadequate liver, kidney, and blood test results
* Received any investigational drug or device within the past 30 days or plans to during the study period
* Has reproductive potential and does not agree to take proper contraceptive measures
* Has active cancer requiring chemotherapy/radiation/major surgery within the next 3 months
* Has significant active concurrent medical illness or infection or life expectancy less than 6 months
* In the opinion of the investigator, is unlikely to comply with the protocol or complete the study, has had drug or alcohol dependence within the past year, or has any other condition that might place the participant at increased risk of harm
* Is a participant in the United States after January 2015 with creatinine clearance (CrCL) greater than 95 mL/minute

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2199 (Actual)
Dates: Start 2014-03-25 (Actual); Primary Completion 2016-02-03 (Actual); Study Completion 2016-02-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (228):
- United States (28):
  - Phoenix, Arizona
  - Escondido, California
  - Newport Beach, California
  - Riverside, California
  - San Francisco, California
  - Santa Rosa, California
  - Denver, Colorado
  - Stamford, Connecticut
  - Newark, Delaware
  - Clearwater, Florida
  - Daytona Beach, Florida
  - Jupiter, Florida
  - Rockledge, Florida
  - Sarasota, Florida
  - Tampa, Florida
  - Boise, Idaho
  - Auburn, Maine
  - Rochester, Minnesota
  - Allentown, Pennsylvania
  - Butler, Pennsylvania
  - Camp Hill, Pennsylvania
  - Hershey, Pennsylvania
  - Jackson, Tennessee
  - Dallas, Texas
  - Fort Worth, Texas
  - Plano, Texas
  - Tyler, Texas
  - Richmond, Virginia
- Austria (5):
  - Graz
  - Innsbruck
  - Linz
  - Mödling
  - Vienna
- Belgium (10):
  - Brussels
  - Genk
  - Ghent
  - Hasselt
  - Huy
  - Leuven
  - Liège
  - Mechelen
  - Tienen
  - Turnhout
- Bulgaria (9):
  - Burgas
  - Gabrovo
  - Pazardzhik
  - Pleven
  - Plovdiv
  - Sofia
  - Stara Zagora
  - Varna
  - Veliko Tarnovo
- Czechia (10):
  - Brno
  - Český Krumlov
  - Havlíčkův Brod
  - Hodonín
  - Kolín
  - Kroměříž
  - Náchod
  - Prague
  - Příbram
  - Slaný
- Denmark (13):
  - Aalborg
  - First site in, Copenhagen
  - Second site in, Copenhagen
  - Frederiksberg
  - Hellerup
  - Herning
  - Holbæk
  - Køge
  - Silkeborg
  - Slagelse
  - Svendborg
  - Vejle
  - Viborg
- France (15):
  - Angers
  - Bordeaux
  - Bron
  - Corbeil-Essonnes
  - Dijon
  - Grenoble
  - Lyon
  - Marseille
  - Montfermeil
  - Montpellier
  - Nice
  - Paris
  - Saint-Denis
  - Toulouse
  - Vandœuvre-lès-Nancy
- Germany (20):
  - Bad Berka
  - Berlin
  - Bielefeld
  - Coburg
  - Dortmund
  - Dresden
  - Freiburg im Breisgau
  - Giessen
  - Hamburg
  - Heidelberg
  - Bad Friedrichshall, Heilbronn
  - Langen
  - Leipzig
  - Ludwigsburg
  - Mainz
  - Marburg
  - Mönchengladbach
  - München
  - Paderborn
  - Regensburg
- Hungary (16):
  - Balatonfüred
  - First site in, Budapest
  - Second site in, Budapest
  - Cegléd
  - Debrecen
  - Győr
  - Gyula
  - Hódmezővásárhely
  - Kecskemét
  - Nagykanizsa
  - Pécs
  - Szeged
  - Székesfehérvár
  - Szolnok
  - Szombathely
  - Zalaegerszeg
- Israel (9):
  - Afula
  - Ashkelon
  - Hadera
  - Haifa
  - Holon
  - Jerusalem
  - Kfar Saba
  - Ramat Gan
  - Tel Aviv
- Italy (11):
  - Acquaviva delle Fonti, BA
  - Santa Maria Capua Vetere, CE
  - Mestre, VE
  - Bologna
  - Catania
  - Chieti
  - Napoli
  - Pavia
  - First site in, Roma
  - Second site in, Roma
  - Trieste
- Netherlands (7):
  - Amsterdam
  - Hilversum
  - Leeuwarden
  - Rotterdam
  - The Hague
  - Venlo
  - Zwolle
- Poland (8):
  - Elblag
  - Krakow
  - Lodz
  - Lublin
  - Puławy
  - Torun
  - Warsaw
  - Wroclaw
- Romania (12):
  - Oradea, Bihor County
  - Craiova, Dolj
  - Focşani, Vrancea
  - Baia Mare
  - Brăila
  - Bucharest
  - Cluj-Napoca
  - Iași
  - Piteşti
  - Târgovişte
  - Târgu Mureş
  - Timișoara
- Russia (7):
  - Barnaul
  - Kemerovo
  - Moscow
  - Novosibirsk
  - Saint Petersburg
  - Tyumen
  - Yaroslavl
- Spain (15):
  - Sant Joan d'Alacant, Alicante
  - Sabadell, Barcelona
  - Salt, Girona
  - Almería
  - First site in, Barcelona
  - Second site in, Barcelona
  - Granada
  - Lugo
  - First site in, Madrid
  - Second site in, Madrid
  - Third site in, Madrid
  - Ourense
  - Santiago de Compostela
  - Valencia
  - Vigo
- Sweden (2):
  - Helsingborg
  - Uppsala
- Ukraine (9):
  - Cherkasy
  - Ivano-Frankivsk
  - Kharkiv
  - Kyiv
  - Odesa
  - Uzhhorod
  - Vinnytsia
  - Zaporizhzhia
  - Zhytomyr
- United Kingdom (22):
  - Romford, Essex
  - Southampton, Hampshire
  - Blackpool, Lancashire
  - Barnet
  - Basildon
  - Birmingham
  - Bournemouth
  - Bradford
  - Chertsey
  - Doncaster
  - Dundee
  - Harrow
  - Leeds
  - Leicester
  - Liverpool
  - Llanelli
  - London
  - Luton
  - Newport
  - Oxford
  - Plymouth
  - Swansea

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

REFERENCES:
- [Background] Giugliano RP, Ruff CT, Braunwald E, Murphy SA, Wiviott SD, Halperin JL, Waldo AL, Ezekowitz MD, Weitz JI, Spinar J, Ruzyllo W, Ruda M, Koretsune Y, Betcher J, Shi M, Grip LT, Patel SP, Patel I, Hanyok JJ, Mercuri M, Antman EM; ENGAGE AF-TIMI 48 Investigators. Edoxaban versus warfarin in patients with atrial fibrillation. N Engl J Med. 2013 Nov 28;369(22):2093-104. doi: 10.1056/NEJMoa1310907. Epub 2013 Nov 19. PMID 24251359
- [Derived] Goette A, Kwong WJ, Ezekowitz MD, Banach M, Hjortshoj SP, Zamoryakhin D, Lip GYH. Edoxaban therapy increases treatment satisfaction and reduces utilization of healthcare resources: an analysis from the EdoxabaN vs. warfarin in subjectS UndeRgoing cardiovErsion of atrial fibrillation (ENSURE-AF) study. Europace. 2018 Dec 1;20(12):1936-1943. doi: 10.1093/europace/euy141. PMID 29947751
- [Derived] Goette A, Merino JL, Ezekowitz MD, Zamoryakhin D, Melino M, Jin J, Mercuri MF, Grosso MA, Fernandez V, Al-Saady N, Pelekh N, Merkely B, Zenin S, Kushnir M, Spinar J, Batushkin V, de Groot JR, Lip GY; ENSURE-AF investigators. Edoxaban versus enoxaparin-warfarin in patients undergoing cardioversion of atrial fibrillation (ENSURE-AF): a randomised, open-label, phase 3b trial. Lancet. 2016 Oct 22;388(10055):1995-2003. doi: 10.1016/S0140-6736(16)31474-X. Epub 2016 Aug 30. PMID 27590218
- [Derived] Lip GY, Merino J, Ezekowitz M, Ellenbogen K, Zamoryakhin D, Lanz H, Jin J, Al-Saadi N, Mercuri M, Goette A. A prospective evaluation of edoxaban compared to warfarin in subjects undergoing cardioversion of atrial fibrillation: The EdoxabaN vs. warfarin in subjectS UndeRgoing cardiovErsion of Atrial Fibrillation (ENSURE-AF) study. Am Heart J. 2015 May;169(5):597-604.e5. doi: 10.1016/j.ahj.2015.02.009. Epub 2015 Feb 21. PMID 25965706

RESULTS

PARTICIPANT FLOW:
Groups:
- Edoxaban: Participants randomized to receive Edoxaban
- Warfarin: Participants randomized to receive Warfarin
Period: Overall Study
Arm/Group | Edoxaban | Warfarin
Started | 1095 | 1104
Intent to Treat Analysis Set | 1095 | 1104
Received Study Drug | 1067 | 1082
Safety Analysis Set | 1067 | 1082
Completed | 1041 | 1014
Not Completed | 54 | 90
Not completed — Protocol Violation | 10 | 9
Not completed — Physician Decision | 5 | 10
Not completed — Adverse event, serious fatal | 1 | 6
Not completed — Adverse Event | 7 | 6
Not completed — Withdrawal by Subject | 17 | 29
Not completed — Other | 14 | 29
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Edoxaban | Warfarin | Total
Number analyzed (Participants) | 1095 | 1104 | 2199
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.3 (10.34) | 64.2 (10.75) | 64.2 (10.54)
Age, Customized [Count of Participants; unit: Participants]
  Age, Categorical: <75 years | 923 | 917 | 1840
  Age, Categorical: ≥75 years | 172 | 187 | 359
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 374 | 382 | 756
  Male | 721 | 722 | 1443
Region of Enrollment [Number; unit: participants]
  Romania | 68 | 54 | 122
  Hungary | 89 | 90 | 179
  United States | 46 | 49 | 95
  Czechia | 86 | 87 | 173
  Ukraine | 206 | 224 | 430
  United Kingdom | 76 | 83 | 159
  Russia | 110 | 106 | 216
  Spain | 73 | 69 | 142
  Austria | 19 | 13 | 32
  Netherlands | 24 | 23 | 47
  Sweden | 7 | 7 | 14
  Belgium | 19 | 22 | 41
  Denmark | 26 | 31 | 57
  Poland | 21 | 33 | 54
  Italy | 34 | 35 | 69
  Israel | 39 | 43 | 82
  Bulgaria | 70 | 55 | 125
  France | 26 | 13 | 39
  Germany | 56 | 67 | 123

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Composite Endpoint of Stroke, Systemic Embolic Stroke (SEE), Myocardial Infarction (MI) and Cardiovascular (CV) Mortality From Randomization to End of Follow up
Time Frame: Randomization to end of follow-up (within 2 years)
Population: This outcome was assessed in the Intent-to-Treat (ITT) Analysis Set.
Measure: Number; unit: Percentage of participants
Arm/Group | Edoxaban | Warfarin
Number analyzed (Participants) | 1095 | 1104
Percentage of participants | 0.5 | 1
Statistical Analysis 1: Comparison: Edoxaban vs Warfarin; Test type: Other; Odds Ratio (OR) = 0.46, 95% CI 2-sided [0.12 to 1.43]

2. Primary Outcome: Percentage of Participants With Composite Endpoints of Major and Clinically-relevant Non-major (CRNM) Bleeding
Time Frame: During treatment period (within 2 years)
Population: This outcome was assessed in the Safety Analysis Set.
Measure: Number; unit: Percentage of participants
Arm/Group | Edoxaban | Warfarin
Number analyzed (Participants) | 1067 | 1082
Percentage of participants | 1.5 | 1
Statistical Analysis 1: Comparison: Edoxaban vs Warfarin; Test type: Other; Odds Ratio (OR) = 1.48, 95% CI 2-sided [0.64 to 3.55]

3. Secondary Outcome: Percentage of Participants With Composite Endpoints of Stroke, SEE, MI, CV Mortality, and Major Bleeding
Time Frame: From randomization to the end of follow-up (within 2 years)
Population: This outcome was assessed in the ITT Analysis Set.
Measure: Number; unit: Percentage of participants
Arm/Group | Edoxaban | Warfarin
Number analyzed (Participants) | 1095 | 1104
Percentage of participants | 0.7 | 1.4
Statistical Analysis 1: Comparison: Edoxaban vs Warfarin; Test type: Other; Difference between percentages = -0.72, 95% CI 2-sided [-1.59 to 0.15]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) were defined as events that started on or after the first dose of study drug or started prior to but then became worse after the first dose of study drug through 30 days after the last dose of study drug (within 2 years).
Description: This table includes counts of participants in the Safety Analysis Set. Participants who experienced more than one episode of an adverse event are counted only once within a preferred term. Participants who experienced more than one adverse event within a system organ class are counted once for each preferred term, but only once for the system organ class.
Arm/Group | Edoxaban | Warfarin
All-Cause Mortality (participants affected / at risk) | 1/1067 | 5/1082
Serious Adverse Events (participants affected / at risk) | 85/1067 | 83/1082
Other Adverse Events (participants affected / at risk) | 53/1067 | 53/1082
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Edoxaban (N=1067) | Warfarin (N=1082)
Hypertensive crisis (Vascular disorders) | 1 (1) | 1 (1)
Aortic aneurysm rupture (Vascular disorders) | 0 (0) | 1 (1) — Aneurysm with rupture abdominal aorta
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Haemodynamic instability (Vascular disorders) | 1 (1) | 0 (0)
Peripheral artery thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Peripheral embolism (Vascular disorders) | 1 (1) | 0 (0)
Thrombophlebitis (Vascular disorders) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 1 (1)
Death (General disorders) | 0 (0) | 1 (1)
Drug effect increased (General disorders) | 0 (0) | 1 (1)
Injection site bruising (General disorders) | 1 (1) | 0 (0)
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Traumatic haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
International normalised ratio increased (Investigations) | 4 (4) | 10 (10)
Liver function test abnormal (Investigations) | 2 (2) | 1 (1)
Blood urine present (Investigations) | 1 (1) | 0 (0)
Coagulation test abnormal (Investigations) | 0 (0) | 1 (1)
International normalised ratio fluctuation (Investigations) | 0 (0) | 1 (1)
Oxygen saturation decreased (Investigations) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 20 (20) | 14 (14)
Cardiac failure (Cardiac disorders) | 3 (3) | 6 (6) — Decompensated heart failure
Cardiac failure congestive (Cardiac disorders) | 5 (5) | 3 (3) — Acute, congestive heart failure
Atrial flutter (Cardiac disorders) | 3 (3) | 2 (2)
Sick sinus syndrome (Cardiac disorders) | 2 (2) | 2 (2)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 2 (2)
Bradycardia (Cardiac disorders) | 2 (2) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 3 (3) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 2 (2) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 2 (2)
Palpitations (Cardiac disorders) | 2 (2) | 1 (1)
Angina unstable (Cardiac disorders) | 0 (0) | 2 (2)
Atrioventricular block complete (Cardiac disorders) | 2 (2) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 2 (2) — Cardiac arrest, ventricular fibrillation
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Atrioventricular block second degree (Cardiac disorders) | 0 (0) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0)
Chordae tendinae rupture (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Left ventricular failure (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Torsade de pointes (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Mediastinal cyst (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulomonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Hypocoagulable state (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 2 (2)
Syncope (Nervous system disorders) | 2 (2) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Loss of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 0 (0) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Retroperitoneal haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Spigelian hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 3 (3) | 2 (2)
Haematuria (Renal and urinary disorders) | 1 (1) | 1 (1)
Cystitis haemorrhagic (Renal and urinary disorders) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Hyperadrenocorticism (Endocrine disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 4 (4) | 4 (4)
Erysipelas (Infections and infestations) | 1 (1) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Arthritis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Chronic sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 0 (0)
Endocarditis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Infective aneurysm (Infections and infestations) | 1 (1) | 0 (0)
Liver abscess (Infections and infestations) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia haemophilus (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Edoxaban (N=1067) | Warfarin (N=1082)
Atrial fibrillation (Cardiac disorders) | 53 (53) | 53 (53)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days